CLINICAL TRIAL: NCT07023250
Title: Sensorineural Hearing Loss Imprint on Manual Dexterity and Coordination: Pediatric and Adolescent Innovative Study
Brief Title: Sensorineural Hearing Loss Imprint
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor, Cairo University
Other Study IDs: Sensorineural Hearing Loss
Record Dates: First submitted 2025-06-04; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sensorineural Hearing Loss Pediatric and Adolescent
  Interventions: Other: manual dexterity and coordination skills
- normal group
  Interventions: Other: manual dexterity and coordination skills

INTERVENTIONS:
Other: manual dexterity and coordination skills — The outcomes were assessed by the use of Bruininks-Oseretsky Test scale of motor proficiency (BOT-2) subtests (3,4&7) for Manual Dexterity, Bilateral Coordination and Upper Limb Coordination respectively. The Bruininks-Oseretsky Examination of Motor Proficiency, Second Edition, evaluates motor performance in various areas such as Manual Dexterity, Bilateral Coordination and Upper Limb Coordination.
  It utilizes subtests and complex structures to diagnose developmental and coordination issues among individuals aged four to twenty-one years old. The test is norm-referenced and purpose-oriented to assess motor abilities. The reliability and validity of the test were 0.78 and 0.84, respectively (Kosari et al., 2013; Ebrahimi et al., 2017; Yassin et al., 2020).

SUMMARY:
this study will investigate the consequences of sensorineural hearing loss on manual dexterity and coordination skills in Children.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with a clinical diagnosis of severe to profound SNHL only. Their ages were between ten to sixteen years, able to understand simple instructions by sign language, able to use both upper and lower limbs, walk and practice daily living activities independently.

Exclusion Criteria:

* Children with cochlear implantation, any cognitive, physical, visual, or neurological conditions (other than SNHI and vestibular impairment), history of previous upper, lower limbs, trunk deformity or surgery. All of these cases were confirmed by medical records and examined by a Physical therapist, Pediatrician, and Audiologist

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Forty-five children from both genders and their ages ranged from ten to sixteen years old were recruited from Public School for the Deaf and Hard of Hearing in Banimazar district, Minia Governorate, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
manual dexterity and coordination | it will be measured only one time in evaluation

IPD SHARING:
Plan to Share IPD: Undecided